CLINICAL TRIAL: NCT02592902
Title: Recurrent Respiratory Papillomatosis and Extraesophageal Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ENT-papilomatosis
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Recurrent Respiratory Papillomatosis; Extra Oesophageal Reflux; Laryngeal Cyst
Keywords: recurrent respiratory papillomatosis; extra oesophageal reflux; laryngeal cyst; phonosurgery; oesophageal impedance
MeSH Terms: conditions — Recurrent respiratory papillomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recurrent respiratory papillomatosis (Active Comparator): Patients with recurrent respiratory papillomatosis (RRP) - surgical collection of histology specimen from the vocal cords and rear laryngeal commissure, performance of immunohistochemical analysis - proof of pepsin, HPV 6 and 11, herpes simplex virus (HSV) type 2, chlamydia trachomasis, and assessment of the dysplasia.
  Interventions: Procedure: Surgical collection of histology specimen; Procedure: Performance of immunohistochemical analysis
- Laryngeal cyst - control group (Active Comparator): Patients with laryngeal cyst - surgical collection of a histology specimen from the vocal cords and rear laryngeal commissure, performance of immunohistochemical analysis - proof of pepsin and HPV 6 and 11, herpes simplex virus (HSV) type 2 and chlamydia trachomasis.
  Interventions: Procedure: Surgical collection of histology specimen; Procedure: Performance of immunohistochemical analysis

INTERVENTIONS:
Procedure: Surgical collection of histology specimen — Collection of a histology specimen from the vocal cords and rear laryngeal commissure
Procedure: Performance of immunohistochemical analysis — Immunohistochemical analysis - presence of pepsin, HPV 6 and 11, HSV 2 and chlamydia trachomasis

SUMMARY:
The purpose of the study was to determine, whether patients with recurrent respiratory papillomatosis (RRP) suffer from extra oesophageal reflux more often than patients with laryngeal cyst (control group).

DETAILED DESCRIPTION:
Recurrent respiratory papillomatosis (RRP) is a chronic viral disease, which affects children and adults as well. It is characterised by grow of squamous cell tumours on mucosa of aerodigestive tract, with predilection for the larynx. The disease is caused by the human papillomavirus (HPV). However, in contrast to the low incidence of RRP, HPV prevalence is common. It is indicated that other factors may contribute to the pathogenesis of RRP. One such factor might be extraesophageal reflux (EER). We investigated whether patients with RRP suffer more often from EER.

ELIGIBILITY:
Inclusion Criteria:

* age 1-75 years
* cooperating patients with laryngeal papillomatosis
* patients tolerating impedance probe
* signed informed consent, consent with the examinations
* control group of patients with a cyst or vocal cord polyp (reflux finding score 0-2) and/or patients indicated to augmentation, medialization or lateralization of the vocal cords

Exclusion Criteria:

* patients non-tolerating impedance catheter
* patients who do not understand Czech language
* patients who do not proclaim consent with enrolment into the study
* patients who do not proclaim consent with the planned examinations
* patients after surgical treatment of tumour of the swallowing or respiratory tract

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of EER (percentage) | 36 months
  The occurrence of extra oesophageal reflux will be assessed in both study groups.

SECONDARY OUTCOMES:
Presence of pepsin | 36 months
  The presence of pepsin (yes-no) will be assessed in both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Formanek, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Czech Republic, Czechia

REFERENCES:
- [Background] Derkay CS, Wiatrak B. Recurrent respiratory papillomatosis: a review. Laryngoscope. 2008 Jul;118(7):1236-47. doi: 10.1097/MLG.0b013e31816a7135. PMID 18496162
- [Background] Gallagher TQ, Derkay CS. Recurrent respiratory papillomatosis: update 2008. Curr Opin Otolaryngol Head Neck Surg. 2008 Dec;16(6):536-42. doi: 10.1097/MOO.0b013e328316930e. PMID 19005325
- [Background] Gallagher TQ, Derkay CS. Pharmacotherapy of recurrent respiratory papillomatosis: an expert opinion. Expert Opin Pharmacother. 2009 Mar;10(4):645-55. doi: 10.1517/14656560902793530. PMID 19284366
- [Background] Goon P, Sonnex C, Jani P, Stanley M, Sudhoff H. Recurrent respiratory papillomatosis: an overview of current thinking and treatment. Eur Arch Otorhinolaryngol. 2008 Feb;265(2):147-51. doi: 10.1007/s00405-007-0546-z. Epub 2007 Nov 29. PMID 18046565
- [Background] Kashima HK, Shah F, Lyles A, Glackin R, Muhammad N, Turner L, Van Zandt S, Whitt S, Shah K. A comparison of risk factors in juvenile-onset and adult-onset recurrent respiratory papillomatosis. Laryngoscope. 1992 Jan;102(1):9-13. doi: 10.1288/00005537-199201000-00002. PMID 1309932
- [Background] Maloney EM, Unger ER, Tucker RA, Swan D, Karem K, Todd NW, Reeves WC. Longitudinal measures of human papillomavirus 6 and 11 viral loads and antibody response in children with recurrent respiratory papillomatosis. Arch Otolaryngol Head Neck Surg. 2006 Jul;132(7):711-5. doi: 10.1001/archotol.132.7.711. PMID 16847177
- [Background] Mammas IN, Sourvinos G, Spandidos DA. Human papilloma virus (HPV) infection in children and adolescents. Eur J Pediatr. 2009 Mar;168(3):267-73. doi: 10.1007/s00431-008-0882-z. Epub 2008 Dec 3. PMID 19050916
- [Background] McKenna M, Brodsky L. Extraesophageal acid reflux and recurrent respiratory papilloma in children. Int J Pediatr Otorhinolaryngol. 2005 May;69(5):597-605. doi: 10.1016/j.ijporl.2004.11.021. PMID 15850681